CLINICAL TRIAL: NCT01943474
Title: The AccuCath Intravenous Catheter System With Retractable Coiled Tip Guidewire and Conventional Peripheral Intravenous Catheters: A Prospective, Randomized, Controlled Comparison by General Hospital Nursing Staff
Brief Title: AccuCath Guidewire Intravenous (IV) Device Versus Conventional IV Catheter In General Nursing Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDVP-001/VPW-STP-00004
Record Dates: First submitted 2013-04-08; First posted 2013-09-17 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Vascular Access Complication
Keywords: IV Catheter comparison; AccuCath versus Conventional IV Catheters; IV Catheter Study; IV Catheter User Preference Comparison; First Attempt Success Rate for IV Catheters; AccuCath Device Performance; Complication Rates for IV Catheters; Average Dwell Time for IV Catheters; Patient Satisfaction with IV Catheters; Clinician Satisfaction with AccuCath Device Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AccuCath IV Catheter Device (Experimental): AccuCath IV Catheter System will be used for IV therapy during inpatient stay. Intervention includes vascular access, fluid infusion, and blood sample removal
  Interventions: Device: AccuCath IV Catheter Device
- Conventional IV Catheter Device (Active Comparator): Conventional IV catheter (current catheter) will be used for IV therapy during inpatient stay. Intervention includes vascular access, fluid infusion, and blood sample removal
  Interventions: Device: Conventional IV Catheter Device

INTERVENTIONS:
Device: AccuCath IV Catheter Device — Vascular access and indwelling catheter placement via study device for infusion of fluids and removal of blood samples.
  Other Names: Rapid Intravascular Start System (RIVS); AccuCath System; AccuCath IV device; AccuCath; AccuCath PIV; AccuCath Short IV; AccuCath IV Catheter
  Arms: AccuCath IV Catheter Device
Device: Conventional IV Catheter Device — Vascular access and indwelling catheter placement via control device for infusion of fluids and removal of blood samples.
  Other Names: Insyte Autoguard; Insyte Autoguard PIV; Insyte Autoguard IV Catheter; Insyte Autoguard IV device
  Arms: Conventional IV Catheter Device

SUMMARY:
The study will test a hypothesis that the AccuCath™ System will have a higher rate of successful first attempt peripheral intravenous (IV) placement, higher completion of therapy, fewer complications, longer dwell times, and higher user satisfaction compared to conventional IV catheters.

DETAILED DESCRIPTION:
This study is designed to evaluate user/physician preference as it relates to use of a 510(k) cleared vascular access and catheter device compared with conventional needle/catheter vascular access devices, in terms of first stick success rates, dwell time, device-related vascular complications and adverse events and overall user and patient satisfaction. As noted above, the study is designed to formally test the hypothesis that the AccuCath™ System will exhibit superiority in terms of the rate of successful first attempt peripheral IV placement, higher completion of therapy, fewer complications, longer dwell times and higher user satisfaction compared to conventional intravenous catheters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years or ≤ 89 years old;
2. Capable and willing to give informed consent;
3. English speaking;
4. Acceptable candidate for an elective, non-emergent peripheral intravenous (PIV) catheter placement as determined by ordering physician;
5. Admitted to study inpatient unit.

Exclusion Criteria:

1. Male or female, < 18 years old or > 89 years old;
2. Requirement for emergent IV placement (patient's condition would be compromised if there is a delay in IV placement);
3. Previous venous grafts or surgery at the target vessel access site;
4. Currently involved in other investigational clinical trials (unless permission is granted by other study principal investigator [PI]);
5. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Rowbottom, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Bette Idemoto, PhD, RN, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional IV Catheter Device: Conventional IV catheter (current catheter) will be used for IV therapy during inpatient stay. Interventions include vascular access, administration of fluids, and removal of blood samples.
  Conventional IV Catheter Device: Vascular access and indwelling catheter placement via control device for infusion of fluids and removal of blood samples.
Period: Overall Study
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Started | 123 | 125
Completed | 123 | 125
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device | Total
Number analyzed (Participants) | 123 | 125 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (15.5) | 62.2 (14.5) | 62.5 (15)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 69 | 127
  >=65 years | 65 | 56 | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 69 | 118
  Male | 74 | 56 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 54 | 103
  White | 73 | 67 | 140
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 123 | 123 | 246
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 123 | 125 | 248

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rate With Peripheral IV Catheter Placement
Description: The primary outcomes measure is to observe first attempt success rate in patients requiring peripheral IV access by documenting the number of catheter attempts (each new catheter) required to complete successful peripheral IV placement.
Time Frame: At catheter placement, an expected average of 10 minutes
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Number analyzed (Participants) | 123 | 125
percentage of participants | 89 [82.8 to 93.7] | 47 [38.7 to 55.9]
Statistical Analysis 1: Comparison: AccuCath IV Catheter Device vs Conventional IV Catheter Device; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Secondary Outcome: Completion of IV Therapy
Description: Completion of IV therapy will measure whether the catheter remained in place for the duration of required intravenous treatment during the inpatient stay (~ up to 7 days).
Time Frame: Study exit/At catheter removal (~ up to 7 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Number analyzed (Participants) | 123 | 125
percentage of participants | 89.4 [82.8 to 93.7] | 34.4 [26.6 to 43.1]
Statistical Analysis 1: Comparison: AccuCath IV Catheter Device vs Conventional IV Catheter Device; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Secondary Outcome: Complications of Peripheral IV Therapy
Description: Will measure the rate of observed (anticipated) complications of IV therapy - infection, occlusion, infiltration, extravasation, phlebitis, dislodgement, leaking/bleeding at site, patient complaints of pain without other identifiable cause, and other (~ up to 7 days).
Time Frame: From during to post IV catheter placement up to study exit (~ up to 7 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Number analyzed (Participants) | 123 | 125
percentage of participants | 8 [4.5 to 14.3] | 52 [43.3 to 60.6]
Statistical Analysis 1: Comparison: AccuCath IV Catheter Device vs Conventional IV Catheter Device; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Secondary Outcome: Catheter Dwell Time
Description: Will measure total catheter dwell time to the nearest hour (total time in hours for functioning catheter) ~ up to 7 days.
Time Frame: Study Exit/At catheter removal (~ up to 7 days)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Number analyzed (Participants) | 123 | 125
hours | 105 (61) | 35 (25)
Statistical Analysis 1: Comparison: AccuCath IV Catheter Device vs Conventional IV Catheter Device; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Patient Satisfaction At Insertion
Description: Will survey patients regarding satisfaction with catheter insertion using a 5-point Likert scale. 5 - Very satisfied, 4 - Somewhat satisfied, 3 - Neutral, 2 - Somewhat unsatisfied, 1 - Very unsatisfied. 3 and above are considered positive. 2 and below are considered negative.
Time Frame: At catheter insertion, initial 3-15 minutes after insertion procedure completed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Number analyzed (Participants) | 123 | 125
units on a scale | 4.6 (0.69) | 3.0 (1.27)
Statistical Analysis 1: Comparison: AccuCath IV Catheter Device vs Conventional IV Catheter Device; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Clinician Satisfaction
Description: Will measure clinician satisfaction of the AccuCath IV device via a 5 point Likert scale survey based on overall catheter performance during experience and use. 5 - Very satisfied, 4 - Somewhat satisfied, 3 - Neutral, 2 - Somewhat unsatisfied, 1 - Very unsatisfied. 3 and above are considered positive. 2 and below are considered negative.
Time Frame: At completion of study after all patients have been enrolled (approximately 6 months from study initiation)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | AccuCath IV Catheter Device
Number analyzed (Participants) | 18
units on a scale | 4 [1 to 5]

7. Secondary Outcome: Adverse Events
Description: Will measure the number and severity of adverse events associated with peripheral IV initiation and indwelling catheter time (anticipated to be similar in both groups). This period will generally include up to 7 days of total IV dwell time.
Time Frame: During and post IV catheter placement until study exit (maximum of 6 months).
Measure: Number; unit: percentage of participants
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Number analyzed (Participants) | 123 | 125
percentage of participants
  Infiltration | 2.4 | 26.4
  Phlebitis | 0.8 | 8.8
  Leaking | 0.8 | 5.6
  Occlusion | 1.6 | 5.6
  Dislodgement | 2.4 | 4.8

8. Secondary Outcome: Patient Satisfaction Comfort Comparison
Description: Patient satisfaction with comfort of IV insertion compared to most recent previous IV insertion using a 5-point Likert scale. 5 - Very satisfied, 4 - Somewhat satisfied, 3 - Neutral, 2 - Somewhat unsatisfied, 1 - Very unsatisfied. 3 and above are considered positive. 2 and below are considered negative.
Time Frame: Immediately after catheter insertion, within the first 3-15 minutes of insertion procedure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Number analyzed (Participants) | 123 | 125
units on a scale | 4.2 (1.02) | 2.86 (1.18)
Statistical Analysis 1: Comparison: AccuCath IV Catheter Device vs Conventional IV Catheter Device; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

9. Secondary Outcome: Patient Satisfaction With Overall IV Performance
Description: Patient satisfaction with overall IV performance at IV removal using a 5-point Likert scale. 5 - Very satisfied, 4 - Somewhat satisfied, 3 - Neutral, 2 - Somewhat unsatisfied, 1 - Very unsatisfied. 3 and above are considered positive. 2 and below are considered negative.
Time Frame: At IV removal (usually after 1-7 days of IV dwell time)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Number analyzed (Participants) | 123 | 125
units on a scale | 4.84 (0.41) | 2.84 (1.01)
Statistical Analysis 1: Comparison: AccuCath IV Catheter Device vs Conventional IV Catheter Device; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During study enrollment from April 2013 - June 2013
Description: Adverse events are the anticipated complications of IV therapy.
Arm/Group | AccuCath IV Catheter Device | Conventional IV Catheter Device
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/125
Other Adverse Events (participants affected / at risk) | 10/123 | 65/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AccuCath IV Catheter Device (N=123) | Conventional IV Catheter Device (N=125)
Phlebitis (Vascular disorders) | 1 | 11
Infiltration (Vascular disorders) | 3 | 33
Dislodgement (Vascular disorders) | 3 | 6
Occlusion (Vascular disorders) | 2 | 7
Leaking (Vascular disorders) | 1 | 7
Infection (Infections and infestations) | 0 | 1
Pain (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less